CLINICAL TRIAL: NCT03955458
Title: A Phase-4, Multicenter, Randomized, Active-Controlled Study to Evaluate the Efficacy and Safety of EXPAREL When Administered Via Fascia Iliaca Compartment Block Versus Fascia Iliaca Compartment Block With Continuous Infusion of Ropivacaine Per Standard of Care Through a Catheter in Intertrochanteric Hip Fracture Patients
Brief Title: EXPAREL Facia Iliaca Compartment Block for Intertrochanteric Hip Fracture
Acronym: RESTORE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-415
Record Dates: First submitted 2019-05-14; First posted 2019-05-20 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Hip Fractures; Intertrochanteric Fractures
Keywords: EXPAREL; FICB; Fascia Iliaca Compartment Block; Ropivacaine
MeSH Terms: conditions — Hip Fractures | interventions — Ropivacaine; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FICB with EXPAREL (Experimental): Group 1: Suprainguinal Fascia Iliaca Compartment Block (FICB) with EXPAREL and bupivacaine HCl
  Interventions: Drug: EXPAREL; Drug: Bupivacaine Hydrochloride
- FICB with Standard of Care: ropivacaine (Active Comparator): Suprainguinal FICB with continuous infusion of local anesthetic (ropivacaine) via catheter placed in the FIC.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: EXPAREL — FICB with EXPAREL + Bupivacaine HCL (single dose)
  Arms: FICB with EXPAREL
Drug: Ropivacaine — FICB with continuous infusion of ropivacaine
  Arms: FICB with Standard of Care: ropivacaine
Drug: Bupivacaine Hydrochloride — FICB with EXPAREL + Bupivacaine HCL (Single dose)
  Arms: FICB with EXPAREL

SUMMARY:
This study evaluates the effect of EXPAREL on total opioid consumption through 72 hours following fascia iliaca compartment block (FICB) in subjects undergoing repair of intertrochanteric hip fracture.

DETAILED DESCRIPTION:
The current standard of care treatment for pain relief in patients with intertrochanteric hip fracture is a FICB with continuous infusion of ropivacaine given via catheter.

In this study, some people will receive a single injection FICB with EXPAREL + bupivacaine HCl. The groups will be evaluated to determine the amount of pain medication they took from the FICB to 72 hours after.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between 65 and 85 years of age (inclusive of) at screening.
2. Intertrochanteric femoral fractures with American Society of Anesthesiology physical status 1, 2, or 3.
3. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

1. Hip fracture that requires total arthroplasty.
2. Patients transferred from other hospitals.
3. Patients that have other acute fractures.
4. Pre-existing dementia (Mini-Mental State examination score <20) or delirium (Mini-Mental State examination score <24).
5. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (e.g., amide-type local anesthetics, opioids, bupivacaine, ropivacaine, acetaminophen, NSAIDs).
6. Serious systemic comorbidities that cause a contraindication for EXPAREL/bupivacaine (severe hepatic or renal impairment) or ropivacaine.
7. Use of anticoagulants (including aspirin, except low dose aspirin).
8. Chronic opioid use of ≥ 20 morphine milligram equivalent (MME)/day for more than 7 days in the last 30 days.
9. Body Mass Index (BMI) <17 kg/m2 or >45 kg/m2.
10. Known history of renal or hepatic dysfunction, coagulation or bleeding disorder.
11. Concurrent painful physical condition that may require analgesic treatment (such as long-term, consistent use of opioids) in the post-operative period for pain that is not strictly related to the surgery and which may confound the post-operative assessments based on the physician's discretion.
12. Clinically significant medical disease that, in the opinion of the investigator, would make participation in a clinical study inappropriate. This includes any psychiatric or other conditions that would constitute a contraindication to participation in the study.
13. History of suspected or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
14. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.
15. Previous participation in an EXPAREL study.
16. Resident of a skilled nursing facility (SNF), long-term acute care (LTAC) facility, inpatient rehabilitation facility (IRF), or nursing home. Participants from assisted living facilities will be eligible for the study.

    In addition, the subject may be withdrawn from the study if the subject meets the following criteria during the hospital stay:
17. Any clinically significant event or condition uncovered during the surgery (e.g., excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's post-operative course.
18. Subjects who undergo hip fracture surgery more than 30 hours after admission to the Emergency Department.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Primary objective (total opioid consumption in morphine equivalents) | Through 72 hours post-FICB
  to compare total opioid consumption in morphine equivalents following FICB with EXPAREL +bupivacaine HCl to that following continuous infusion of ropivacaine via catheter, from end of FICB placement through 72 hours post-FICB, in subjects undergoing repair of intertrochanteric hip fracture To be measured as date, time, and dosage of all medication administered from the time ICF is signed to 72-hours post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nayana Nagaraj, MD, PhD, MPH, Study Director — Pacira Biosciences Inc.
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No